CLINICAL TRIAL: NCT02471326
Title: An Exploratory, Open-Label Study of VRC-HIVMAB060-00-AB (VRC01) in Subjects With Chronic HIV Infection Undergoing Analytical Treatment Interruption
Brief Title: VRC-HIVMAB060-00-AB (VRC01) in People With Chronic HIV Infection Undergoing Analytical Treatment Interruption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150140; 15-I-0140 (Other: NIAID IRB)
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: HIV Neutralizing Antibodies; HIV Therapy
MeSH Terms: interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIV Positive Subjects (Experimental): VRC-HIVMAB060-00-AB (VRC01) given in HIV-infected Adults (age 18-65 years) on cART with suppressed viremia
  Interventions: Biological: VRC-HIVMAB060-00-AB (VRC01)

INTERVENTIONS:
Biological: VRC-HIVMAB060-00-AB (VRC01) — A potent HIV-specific monoclonal antibody

SUMMARY:
Background:

- A combination of daily drugs (called cART) can keep human immunodeficiency virus (HIV) very low for a long time. But cART can lose effectiveness and cause permanent side effects. If treatment stops, HIV levels go up again. Researchers want to see if a new product can control HIV levels when a person is off cART.

Objective:

- To see if the new product VRC01 is safe and can control the HIV level in the blood when a person is not taking cART.

Eligibility:

- Adults ages 18-65 with HIV who are willing to interrupt their treatment for at least 24 weeks.

Design:

* Participants will be screened with:
* Physical exam
* Medical history
* Heart tests
* Blood and urine tests.
* Their HIV drugs may be switched. They will keep taking them until a few days after Visit 1.
* Visit 1: Repeat screening procedures.
* Participants will also have genetic testing and leukapheresis. For this, blood will be removed through a needle in one arm and circulated through a machine that removes white blood cells. The rest of the blood is returned through a needle in the other arm.
* They will get the first study drug dose through a thin tube in an arm vein for about 1 hour.
* For 24 weeks, participants will have 16 visits. They will have blood drawn every visit. At some visits they will repeat the screening procedures and get another VRC01 dose. They may have another leukapheresis.
* Four weeks after the last dose, participants will restart their cART. For 20 weeks, they will have monthly visits to repeat the screening procedures and discuss new symptoms.

DETAILED DESCRIPTION:
Recent advances in antibody cloning technologies have led to the discovery of a number of highly potent, HIV-specific, broadly neutralizing monoclonal antibodies from B cells of HIV-infected individuals. It has been shown that certain broadly neutralizing HIV-specific antibodies can prevent acquisition of the virus, suppress viral replication, delay and/or prevent plasma viral rebound following treatment interruption in Simian Immunodeficiency virus (SIV)-infected animals and block cell-to-cell transmission of laboratory-adapted HIV in vitro. However, it is unclear what in vivo effects these antibodies might have on plasma viral rebound in HIV-infected individuals following discontinuation of combination antiretroviral therapy (cART).

In this regard, it has been shown that virtually all infected individuals who initiated cART during the chronic phase of infection experience plasma viral rebound upon cessation of therapy. Current research on the treatment of HIV-infected individuals has been heavily focused on developing strategies aimed at achieving sustained virologic remission in the absence of cART. Thus, it is of great interest to investigate whether a potent HIV-specific monoclonal antibody, such as VRC01, can prevent plasma viral rebound in infected individuals upon discontinuation of cART. We propose to examine the effect of VRC01 on plasma viral rebound in HIV-infected individuals following analytical treatment interruption (ATI).

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Age 18-65 years old.
  2. HIV-1 infection and clinically stable.
  3. In general good health and with an identified primary health care provider for medical management of HIV infection and willing to maintain a relationship with a primary health care provider for medical management of HIV infection while participating in the study.
  4. CD4+ cell count >450 cells/mm^3 at screening.
  5. Documentation of continuous cART treatment with suppression of plasma viral level below the limit of detection for greater than or equal to 3 years. Subjects with blips (i.e., detectable viral levels on cART) prior to screening may be included provided they satisfy the following criteria:

     1. The blips are <400 copies/mL, and
     2. Succeeding viral levels return to levels below the limit of detection on subsequent testing.
  6. Willingness to undergo ATI.
  7. Laboratory values within pre-defined limits at screening:

     1. Absolute neutrophil count >1,000/mm^3.
     2. Hemoglobin levels >10.0 g/dL for men and >9.0 g/dL for women.
     3. Platelet count >100,000/mm^3.
     4. Prothrombin time (PT) and partial thromboplastin time (PTT) <1.5 upper limit of normal (ULN).
     5. Estimated or a measured creatinine clearance rate of greater than or equal to 50 mL/min as determined by the NIH Clinical Center laboratory.
     6. AST and ALT levels of <2.5 x ULN.
  8. Willingness to have samples stored for future research.

Reproductive Risks

Contraception: The effects of VRC01 on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate pregnancy prevention per the investigator. This includes highly reliable established lifestyle of complete abstinence of potentially reproductive sexual activity, or use of BOTH a long term hormonal or barrier (e.g. implant, depot injection, IUD in female participant or female partner of participant) method of contraception that is fully effective prior to dosing, COMBINED WITH a barrier method (male or female condom) for all potentially reproductive sexual activity. Pregnancy prevention must be maintained as effective and practiced continuously for the duration of study participation. Females of childbearing-age must have a negative pregnancy test result prior to receiving VRC01. During the course of the study, if a female participant, or the partner of a male participant suspects or in fact becomes pregnant, the effected participant should inform the study staff immediately, as well as the woman's primary care physician. Subjects must use safe sex practices during the trial, and particularly during the ATI phase, when risk of transmission of HIV may be increased.

* EXCLUSION CRITERIA

  1. Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen (HBsAg), or chronic hepatitis C virus (HCV) infection, as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
  2. Documented virologic failure to >1 cART regimen.
  3. HIV immunotherapy or vaccine(s) received within 1 year prior to screening.
  4. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment.
  5. Receipt of other investigational study agent within 28 days of enrollment.
  6. Any active malignancy that may require systemic chemotherapy or radiation therapy.
  7. Systemic immunosuppressive medications received within 3 months prior to enrollment (Not excluded: corticosteroid nasal spray or inhaler; topical corticosteroids for mild, uncomplicated dermatitis; or oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur [length of therapy less than or equal to 10 days, with completion in greater than or equal to 30 days prior to enrollment]).
  8. History or other clinical evidence of:

     1. Significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction).
     2. Severe illness, malignancy, immunodeficiency other than HIV, or any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study.
  9. Active drug or alcohol use or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.
  10. Breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-13; Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Zhou T, Georgiev I, Wu X, Yang ZY, Dai K, Finzi A, Kwon YD, Scheid JF, Shi W, Xu L, Yang Y, Zhu J, Nussenzweig MC, Sodroski J, Shapiro L, Nabel GJ, Mascola JR, Kwong PD. Structural basis for broad and potent neutralization of HIV-1 by antibody VRC01. Science. 2010 Aug 13;329(5993):811-7. doi: 10.1126/science.1192819. Epub 2010 Jul 8. PMID 20616231
- [Background] Shingai M, Nishimura Y, Klein F, Mouquet H, Donau OK, Plishka R, Buckler-White A, Seaman M, Piatak M Jr, Lifson JD, Dimitrov DS, Nussenzweig MC, Martin MA. Antibody-mediated immunotherapy of macaques chronically infected with SHIV suppresses viraemia. Nature. 2013 Nov 14;503(7475):277-80. doi: 10.1038/nature12746. Epub 2013 Oct 30. PMID 24172896
- [Background] Chun TW, Murray D, Justement JS, Blazkova J, Hallahan CW, Fankuchen O, Gittens K, Benko E, Kovacs C, Moir S, Fauci AS. Broadly neutralizing antibodies suppress HIV in the persistent viral reservoir. Proc Natl Acad Sci U S A. 2014 Sep 9;111(36):13151-6. doi: 10.1073/pnas.1414148111. Epub 2014 Aug 25. PMID 25157148
- [Derived] Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, Salantes DB, Seamon CA, Scheinfeld B, Kwan RW, Learn GH, Proschan MA, Kreider EF, Blazkova J, Bardsley M, Refsland EW, Messer M, Clarridge KE, Tustin NB, Madden PJ, Oden K, O'Dell SJ, Jarocki B, Shiakolas AR, Tressler RL, Doria-Rose NA, Bailer RT, Ledgerwood JE, Capparelli EV, Lynch RM, Graham BS, Moir S, Koup RA, Mascola JR, Hoxie JA, Fauci AS, Tebas P, Chun TW. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med. 2016 Nov 24;375(21):2037-2050. doi: 10.1056/NEJMoa1608243. Epub 2016 Nov 9. PMID 27959728
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0140.html

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Positive Subjects: Drug: VRC-HIVMAB060-00-AB (VRCO1), 40 mg/kg in 100 mL Normal Saline; VRC-HIVMAB060-00-AB (VRCO1) is a potent HIV-specific monoclonal antibody which was given at Baseline, Week 2, and then every 4 weeks for up to a total of 8 doses
Period: Overall Study
Arm/Group | HIV Positive Subjects
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | HIV Positive Subjects
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 or Higher Adverse Events
Description: The primary endpoint was the number of grade 3 or higher adverse events, including serious adverse events, that were possibly related to VRC-HIVMAB060-00-AB (VRCO1).
Time Frame: From the start of the initial infusion until up to 48 weeks.
Population: The analyses included all subjects who received at least one infusion of VRC-HIVMAB060-00-AB (VRCO1).
Measure: Number; unit: Events
Arm/Group | HIV Positive Subjects
Number analyzed (Participants) | 10
Events | 0

2. Secondary Outcome: Subjects Who Met Criteria to Restart Antiretroviral Therapy
Description: The secondary endpoint was the number of subjects who met protocol defined virologic (sustained HIV RNA >1000 copies/mL by Abbott HIV RTPCR at 2 consecutive visits), immunologic (a confirmed >30% decline in CD4 cell count or an absolute CD4 cell count < 350 cells/mm3), or clinical criteria (HIV-related symptoms) to discontinue VRC01 infusions and restart Antiretroviral Therapy (ART).
Time Frame: From Day 3 post initial infusion until up to 28 weeks.
Population: The analyses included all subjects who received at least one infusion of VRC-HIVMAB060-00-AB (VRCO1).
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Positive Subjects
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: up to 48 Weeks
Arm/Group | HIV Positive Subjects
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Positive Subjects (N=10)
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Positive Subjects (N=10)
Nausea (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Influenza like illness (General disorders) | 1
Localised oedema (General disorders) | 1
Diarrhoea infectious (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood calcium decreased (Investigations) | 2
Blood glucose increased (Investigations) | 3
Blood phosphorus decreased (Investigations) | 2
Blood sodium decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02471326/Prot_SAP_000.pdf